CLINICAL TRIAL: NCT06165666
Title: Effectiveness of Physiotherapy for Improving Functionality, Participation and Quality of Life After a Stroke: Single-blind Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Physiotherapy After Stroke
Acronym: EPTAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Concepción Soto-Vidal, Degree Teacher in Physiotherapy, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stroke Project
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: stroke; physiotherapy; clinical trial
MeSH Terms: conditions — Stroke | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned into 2 groups (intervention group (EG) and control group (CG)).
Who Masked: Outcomes Assessor
Masking Description: Single-blind, parallel, randomized controlled clinical trial, allocation ratio 1:1 and with third-party evaluation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (EG) (Experimental): The participants will receive as a therapeutic approach 3 physical therapy sessions/week of 40' duration, for 10 weeks.
  Interventions: Other: Approach by functional objectives
- control group (CG) (Active Comparator): The participants will receive as a therapeutic approach 3 physical therapy sessions/week of 40' duration, for 10 weeks.
  Interventions: Other: Treatment protocol

INTERVENTIONS:
Other: Approach by functional objectives — The therapeutic approach that will be administered to the EG will be based on the training of specific tasks aimed at functional objectives. Each session will begin with activities to activate the muscles of the trunk, pelvis and lower limbs, to modify atypical movement patterns and prepare the muscles for a more effective contraction. Subsequently, activity training will be carried out in a functional and meaningful context, aimed at specific and significant functional objectives for the participant and previously agreed upon with them.
  Arms: intervention group (EG)
Other: Treatment protocol — The therapeutic approach of the participants assigned to the CG will be aimed at maintaining joint ranges and transfer work, passive mobilization of the paretic lower and upper limb, maintenance of sitting posture with/without assistance, transfer from sitting to standing, from standing to sitting. and coordination work. Subsequently, initiation of walking with a support product and/or help, if possible.
  Arms: control group (CG)

SUMMARY:
The World Health Organization (WHO) defines Stroke or Cerebrovascular Accident as clinical sign of focal disorder in brain functioning of rapid onset, with a presumed vascular origin and duration of more than 24 hours. It represents the first cause of physical disability in adults, and approximately half of people who survive stroke present motor and sensitivity disorders, which cause alterations in functionality, especially in activities of daily living, with the consequent impact negative in participation in the environment and the quality of life of people and their families.

The objective of the study is to know the effectiveness of a Physiotherapy intervention, based on the achievement of objectives, in improving functionality, participation and quality of life after a Stroke compared to treatment protocol.

Methodology: single-blind randomized controlled clinical trial. The sample of 62 subjects (31 in each group) will be recruited at the Ramon y Cajal University Hospital. The Physiotherapy intervention will consist of 30 sessions, 3 times/week, for 10 consecutive weeks, in which the treatment for the Experimental Group will be based on training of specific tasks aimed at functional objectives previously agreed upon with the person/user vs. the Control Group who will receive a conventional Physiotherapy treatment protocol. The outcome variables are: perception of quality of life (Spanish version of The Newcastle Stroke-specific Quality of Life Measure); degree of functional disability (Barthel Index); level of gait functionality (Spanish version of Functional Ambulation Categories); dynamic balance and trunk control (Spanish version of Trunk Impairment Scale); postural control (Spanish version of the Postural Assessment Scale for Stroke Patients); and participation in the environment (Spanish version of the Oxford Participation and Activities Questionnaire). They will be collected at three times: before starting the study, initial assessment (V0), at the end of the intervention for each group, intermediate assessment (V1) and 6 months after V0 (V2).

DETAILED DESCRIPTION:
Background:

According to the WHO, stroke represents the first cause of physical disability in the adult population, as well as the second cause of death in industrialized and developed countries, becoming a pathology of great socioeconomic cost. The number of people suffering from stroke, worldwide, has increased considerably in recent decades, especially since the beginning of the global pandemic, presenting itself as a complication of COVID19. In Spain, the incidence of stroke ranges between 150 and 323 cases per 100,000 inhabitants. Its frequency increases with age, especially in the population over 65 years of age, and it is considered that after six months of having suffered a stroke, 26.1% of people die, 41.5% of those affected are independent, and 32.4% have some type of functional dependency.

Among the most frequent sequelae, motor impairment stands out, which is usually considered the main cause of disability in people due to its impact on balance, causing gait disorders and an increased risk of falls, as well as difficulty in handling and performance of activities of daily living (ADL). When these alterations persist over time, they not only hinder functionality but also interfere with the interaction with the environment and the subject's participation in social activities, negatively affecting the perception of their quality of life. This is why Physiotherapy interventions that include training in functional activities are an optimal approach strategy. Recently, based on the International Classification of Functioning, Disability and Health, a paradigm shift is occurring in the treatment of the functionality of people who have suffered a stroke. The European Stroke Organization indicates that during motor recovery, patients learn to optimize their motor, sensory and cognitive functioning through repetitive, goal-oriented, progressive and task-specific training. And here it is worth highlighting the importance of the functional orientation of physiotherapy to help these people maximize health, well-being and quality of life.

Physiotherapy treatment after stroke carries a high cost as it requires specialized personnel in a multidisciplinary team because it is a long-term individualized therapy. Instead of limiting ourselves to teaching compensation methods to recover mobility, motor control and lost balance, it has been proposed to focus on the nervous system's ability to recover previous movement patterns, through functional use and neuroplasticity. Establishing functional goals could be the key to effective decision making, as well as a person-centered outcome measure for Stroke rehabilitation. Based on all this, we consider that the Physiotherapy intervention should be based on the needs of the person instead of pre-established treatment designs.

The latest systematic reviews carried out show that the impact of methodologies based on functionality compared to conventional treatments has not yet been rigorously evaluated. Optimizing physiotherapy treatment would allow us to improve the patient's level of recovery after a stroke, reducing dependency rates and increasing their quality of life, while reducing the number of sessions necessary and the waiting list to access treatment.

Objective:Know the effectiveness of a Physiotherapy intervention, based on the achievement of objectives in improving functionality, participation and quality of life after a Stroke compared to treatment protocol.

Design: Single-blind, parallel, randomized controlled clinical trial, 1:1 allocation ratio and with third-party evaluation. The study has been approved by the Research Ethics Committee of the Ramon y Cajal University Hospital (220/23).

Study population

Inclusion criteria:

* Diagnosis of Stroke between 6 and 24 months before to study access.
* Age ≥ 50 years.
* Signing of the informed consent.

In order to detect differences in functionality, participation and quality of life in favor of the experimental group, a large effect size of d = 0.80, an error α = 0.05 and a power of 90% is assumed. Considering a possible loss to follow-up of 10%, the sample size results in 62 participants.

Methodology: participants are randomly assigned into 2 groups (intervention group (EG) and control group (CG)). All participants will receive as a therapeutic approach 3 sessions/week of 40' duration, for 10 weeks.

The therapeutic approach that will be administered to the EG will be based on the training of specific tasks aimed at functional objectives. Each session will begin with activities to activate the muscles of the trunk, pelvis and lower limbs, to modify atypical movement patterns and prepare the muscles for a more effective contraction. Subsequently, activity training will be carried out in a functional and meaningful context, aimed at specific and significant functional objectives for the participant and previously agreed upon with them. In these sessions, aspects such as postural orientation and stability, movement components and the ability to perform selective movement are taken into account.

The therapeutic approach of the participants assigned to the CG will be aimed at maintaining joint ranges and transfer work, passive mobilization of the paretic lower and upper limb, maintenance of sitting posture with/without assistance, transfer from sitting to standing, from standing to sitting. and coordination work. Subsequently, initiation of walking with a support product and/or help, if possible.

Variables: Perception of quality of life (Spanish version of The Newcastle Stroke-specific Quality of Life Measure. Degree of functional disability (Barthel Index), Functional level of gait (Spanish version of the "Functional Ambulation Categories. Dynamic balance) and trunk control (Spanish version of the Trunk Impairment Scale, Postural control (Spanish version of the Postural Assessment Scale for Stroke and Participation in the environment (Spanish version of the Oxford Participation and Activities Questionnaire. The following will also be collected: age, sex, weight, height, type of stroke, evolution time and most affected hemibody.

Data collection and analysis: data will be collected three times throughout the process: (V0), start of the study; (V1) end of intervention period and (V2), six months after the start of the study. After the measurements (V0, V1 and V2), the data will be analyzed with the Statistical Package for the Social Sciences software, version 25 for Mac.

Descriptive statistics will be performed using means and standard deviations, in the case of quantitative variables with a normal distribution, or medians and interquartile ranges, failing that. Normality will be studied using the Kolmogorov-Smirnov test. For nominal qualitative variables, absolute and relative percentage frequencies will be used.

The homogeneity of descriptive variables and initial outcome variables will be analyzed with the Student t test for independent samples (homoscedastic normal quantitative variables), with the Welch t test (non-heteroscedastic normal quantitative variables) or with the Mann-Whitney U test. (non-normal quantitative variables). In the case of nominal qualitative variables, Pearson's Chi-square test or Fisher's exact test will be used.

To study the differences between the experimental group and the control group, the Student t test for independent samples, the Welch t test or the Mann-Whitney U test will be used.

The database used in the study will be created in the RedCAP system, with the collaboration of the Ramon y Cajal Institute for Health Research Data Science Unit, a secure and structured database that allows open access to information at the institutional level, complying with Open Sciences requirements.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with stroke between 6 and 24 months before the intervention.
* Age 50 or more years.
* Have signed the informed consent.

Exclusion Criteria:

* Present moderate or severe cognitive impairment according to the Pfeiffer Questionnaire.
* Have other serious diseases with a significant impact on functional capacity.
* Suffer previously diagnosed psychiatric pathology.
* Being dependent for activities of daily living before suffering the stroke.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Perception of quality of life | Beginning of the study, end of the therapeutic intervention period and 6 months after the start of the study.
  Spanish version of NewsQoL
Functional disability | Beginning of the study, end of the therapeutic intervention period and 6 months after the start of the study.
  Barthel index
Participation in the environment | Beginning of the study, end of the therapeutic intervention period and 6 months after the start of the study.
  Spanish version Oxford Participation and Activities Questionnaire

SECONDARY OUTCOMES:
Level of gait functionality | Beginning of the study, end of the therapeutic intervention period and 6 months after the start of the study.
  Spanish version of the Functional Ambulation Categories
Dynamic balance and trunk control | Beginning of the study, end of the therapeutic intervention period and 6 months after the start of the study.
  Spanish version of the Trunk Impairment Scale
Postural control | Beginning of the study, end of the therapeutic intervention period and 6 months after the start of the study.
  Spanish version of the Postural Assessment Scale for Stroke Patients

OTHER OUTCOMES:
Cognitive impairment | Prior to inclusion in the study
  Pfeiffer questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Concepción Soto-Vidal, Principal Investigator — University of Alcala
Locations (1):
- Concepción Soto-Vidal, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murie-Fernandez M, Irimia P, Martinez-Vila E, John Meyer M, Teasell R. [Neuro-rehabilitation after stroke]. Neurologia. 2010 Apr;25(3):189-96. Spanish. PMID 20492866
- [Background] Wonsetler EC, Bowden MG. A systematic review of mechanisms of gait speed change post-stroke. Part 2: exercise capacity, muscle activation, kinetics, and kinematics. Top Stroke Rehabil. 2017 Jul;24(5):394-403. doi: 10.1080/10749357.2017.1282413. Epub 2017 Feb 20. PMID 28218021
- [Background] Tan YK, Goh C, Leow AST, Tambyah PA, Ang A, Yap ES, Tu TM, Sharma VK, Yeo LLL, Chan BPL, Tan BYQ. COVID-19 and ischemic stroke: a systematic review and meta-summary of the literature. J Thromb Thrombolysis. 2020 Oct;50(3):587-595. doi: 10.1007/s11239-020-02228-y. PMID 32661757
- [Background] Alessandro L, Olmos LE, Bonamico L, Muzio DM, Ahumada MH, Russo MJ, Allegri RF, Gianella MG, Campora H, Delorme R, Vescovo ME, Lado V, Mastroberti LR, Butus A, Galluzzi HD, Decima G, Ameriso SF. [Multidisciplinary rehabilitation for adult patients with stroke]. Medicina (B Aires). 2020;80(1):54-68. Spanish. PMID 32044742
- [Background] Kwakkel G, Stinear C, Essers B, Munoz-Novoa M, Branscheidt M, Cabanas-Valdes R, Lakicevic S, Lampropoulou S, Luft AR, Marque P, Moore SA, Solomon JM, Swinnen E, Turolla A, Alt Murphy M, Verheyden G. Motor rehabilitation after stroke: European Stroke Organisation (ESO) consensus-based definition and guiding framework. Eur Stroke J. 2023 Dec;8(4):880-894. doi: 10.1177/23969873231191304. Epub 2023 Aug 7. PMID 37548025
- [Background] Leonardi M, Fheodoroff K. Goal Setting with ICF (International Classification of Functioning, Disability and Health) and Multidisciplinary Team Approach in Stroke Rehabilitation. 2021 Jan 15. In: Platz T, editor. Clinical Pathways in Stroke Rehabilitation: Evidence-based Clinical Practice Recommendations [Internet]. Cham (CH): Springer; 2021. Available from http://www.ncbi.nlm.nih.gov/books/NBK585584/ PMID 36315695
- [Background] Rosewilliam S, Roskell CA, Pandyan AD. A systematic review and synthesis of the quantitative and qualitative evidence behind patient-centred goal setting in stroke rehabilitation. Clin Rehabil. 2011 Jun;25(6):501-14. doi: 10.1177/0269215510394467. Epub 2011 Mar 25. PMID 21441308
- [Background] Sugavanam T, Mead G, Bulley C, Donaghy M, van Wijck F. The effects and experiences of goal setting in stroke rehabilitation - a systematic review. Disabil Rehabil. 2013 Feb;35(3):177-90. doi: 10.3109/09638288.2012.690501. Epub 2012 Jun 7. PMID 22671934
- [Result] Azevedo da Costa F, Araujo da Silva DL, da Rocha VM. [The functional condition of patients following a cerebrovascular accident]. Rev Neurol. 2006 May 16-31;42(10):591-5. Spanish. PMID 16703526
- [Derived] Soto-Vidal C, Calvo-Fuente V, Hidalgo-Galante E, Cerezo-Tellez E, Perez-Martin Y, Pacheco-da-Costa S. Effectiveness of Physiotherapy for Improving Functionality, Participation, and Quality of Life after a Stroke: Study Protocol for a Randomized Controlled Clinical Trial. J Pers Med. 2024 Aug 22;14(8):891. doi: 10.3390/jpm14080891. PMID 39202082